CLINICAL TRIAL: NCT07187323
Title: Free Amino-acid Composition of Saliva in Patients With Different Peri-implant and Periodontal Conditions
Brief Title: Free Amino-acid Composition of Peri-implant and Periodontal Conditions
Acronym: AAs
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Lokman Hekim University (Other Government); Ankara University (Other); Ankara Medipol University (Other)
Responsible Party: Principal Investigator, Nur Balci, DDs, PhD, Assoc Prof Dr, Istanbul Medipol University Hospital
Other Study IDs: 645; Istanbul Medipol University (Other: Lokman Hekim University)
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Peri-Implant Health; Peri Implant Mucositis; Peri Implantitis
Keywords: peri-implantitis; amino acids; saliva
MeSH Terms: conditions — Peri-Implantitis | interventions — Sequence Analysis, Protein

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Saliva collection: Saliva and serum sampling Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day.
  The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 10 mL of blood samples were collected by qualified staff from each participant. Saliva and serum were then stored at -80 °C until analysis.
  Interventions: Other: Saliva sampling
- Amino Acid Analysis: Quantitative analysis of amino acids in saliva was carried out using liquid chromatography-tandem mass spectrometry (LC-MS/MS) with a Thermo Scientific TSQ Quantum Access MAX system (Thermo Scientific, Schaumburg, IL, USA).
  Interventions: Other: Amino Acid Analysis

INTERVENTIONS:
Other: Saliva sampling — Unstimulated, whole saliva was collected from all participants across the six study groups following a detailed explanation of the procedure. Initially, individuals were asked to rinse their mouths with filtered water and remain seated in a relaxed position for five minutes. Then, they were instructed to passively drool into a sterile collection tube over a 10-minute period.31 The collected saliva samples were then centrifuged at 3000 ×g for 10 minutes to remove debris and prepare them for storage at -80°C .
  Groups: Saliva collection
Other: Amino Acid Analysis — Saliva samples were deproteinized by mixing with 6% sulfosalicylic acid in a 1:1 ratio, followed by incubation at room temperature for 5 minutes. The mixtures were then centrifuged at 15,000 rpm for 5 minutes. A 10 µL aliquot of the resulting supernatant was diluted with 800 µL of 2 mM tridecafluoroheptanoic acid containing 0.375 M glucosaminic acid and internal standards. The prepared solutions were transferred into autosampler vials for analysis. Calibration standards were generated by combining known concentrations of amino acid standards.
  Groups: Amino Acid Analysis

SUMMARY:
Peri-implant diseases, encompassing peri-implant mucositis and peri-implantitis, are biologically driven inflammatory conditions that threaten the long-term success of dental implants. The microbial signatures and their metabolic products have prompted growing interest in salivary biomarkers, particularly amino acids (AAs), which may reflect both microbial activity and host response.However, despite increasing evidence of periodontal disease, the role of salivary AAs in peri-implant conditions remains underexplored.The aim of this study is to comprehensively evaluate and compare the salivary free amino acid profiles among individuals with peri-implantitis, peri-implant mucositis, and healthy peri-implant mucosa, as well as those with periodontitis, gingivitis, and a healthy periodontium, and seeks to investigate whether distinct salivary amino acid signatures are linked to different stages and types of peri-implant and periodontal inflammation, and to evaluate their potential as non-invasive biomarkers for disease differentiation, activity, and severity

DETAILED DESCRIPTION:
The study included one-hundred and thirty-two patients who applied to the Department of Periodontology at Istanbul Medipol University, Faculty of Dentistry. Four of the one-hundred and thirty-two patients declined to participate in the trial. Two patients were eliminated because they had recently taken antibiotics, six patients were discarded because they had recently received periodontal therapy, and six patients were excluded because they had systemic diseases, resulting in a final sample size of one-hundred and twenty patients .Quantitative analysis of amino acids in saliva was carried out using liquid chromatography-tandem mass spectrometry (LC-MS/MS) with a Thermo Scientific TSQ Quantum Access MAX system.

ELIGIBILITY:
Inclusion Criteria:

* be between 18 and 65 years of age
* have a minimum of 20 natural teeth, excluding third molars (for non-implant-treated groups)
* be edentulous patients treated with implants loaded at least 1 year prior (for implant-treated groups)
* be in a systemically healthy condition.

Exclusion Criteria:

* current tobacco use
* chronic use of any systemic medication
* use of antibiotics, anti-inflammatory drugs (including corticosteroids and NSAIDs), immunosuppressants, beta-blockers, calcium channel blockers, anticoagulants, or hormonal contraceptives within the 3 months prior to the study
* receipt of periodontal therapy within the past 6 months
* pregnancy or breastfeeding
* presence of orthodontic appliances a DMFT index (Decayed, Missing, and Filled Teeth per tooth) greater than 2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients who has healthy implants, the peri implant mucositis patients, peri-implantitis patients, periodontally healthy volunteers, gingivitis and stage 3 grade b patients were enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | 3 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe
Bleeding on probing | 4 months
  Bleeding on probing referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth

SECONDARY OUTCOMES:
saliva analyses for selected molecules | 4 months
  Quantitative analysis of amino acids in saliva was carried out using liquid chromatography-tandem mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No